CLINICAL TRIAL: NCT01387425
Title: Efficacy And Safety Of Smoking Cessation With Varenicline Tartrate In Diabetic Smokers: A Double-Blind, Placebo-Controlled, Randomized, Trial
Brief Title: Efficacy And Safety Of Smoking Cessation With Varenicline Tartrate In Diabetic Smokers: (DIASMOKE)
Acronym: DIASMOKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Catania (Other)
Responsible Party: Principal Investigator, Riccardo Polosa, Professor of Internal Medicine, Universita degli Studi di Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-017599-26
Record Dates: First submitted 2011-06-13; First posted 2011-07-04 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Smoking Cessation; Diabetes
Keywords: Smoking cessation of diabetic smoker
MeSH Terms: conditions — Smoking Cessation; Diabetes Mellitus | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- varenicline (Active Comparator): varenicline 1 mg BID. The duration of active treatment will be 12 weeks.
  Interventions: Drug: varenicline
- control group (Placebo Comparator)
  Interventions: Drug: placebo tablet is made of lactose

INTERVENTIONS:
Drug: varenicline — varenicline at a dose of 1 mg twice a day for 12 week
  Arms: varenicline
Drug: placebo tablet is made of lactose — placebo at a dose of 1 mg twice for 12 week
  Arms: control group

SUMMARY:
Objectives

This protocol is intended to provide information regarding the efficacy and safety of the nicotine partial agonist varenicline tartrate, at a dose of 1 mg twice daily, for smoking cessation in diabetic subjects who smoke. Given that a better understanding of predictors of smoking cessation can be useful in identifying potential quitters and likely relapsers and that little is known about these predictors in diabetics, the role of different predictors of abstinence at the end of the study will also be examined Study Population The study will enroll 150 type 2 diabetic patients (≤ 75 years) who are regular smokers (≥10 cigs/day) and motivated to stop smoking in each of 2 treatment arms (active drug and placebo) Study Design The study is a double-blind, placebo-controlled, randomized clinical trial designed to assess the efficacy and safety of varenicline 1 mg BID in comparison to placebo for smoking cessation. The duration of active treatment will be 12 weeks and subjects will be followed in the nontreatment phase for an additional 12 weeks. This clinical study has an optional research component to prolong the follow up in the nontreatment phase for a full year. Predictors of abstinence at the end of the study will also be examined Study Endpoints Primary Endpoint: Success rates at week 24 in the varenicline vs placebo group. Success rates will be defined as the Continuous Quit Rate since last visit. Subjects will be classified as responders if they are able to maintain abstinence from cigarette smoking during this period of time with end-expiratory exhaled CO measurements ≤ 10 ppm. This measure will be obtained through reports of cigarette use by means of the Nicotine Use Inventory confirmed by a measurement of an end-expiratory exhaled carbon monoxide concentration that is ≤ 10 ppm on the study visit at week 24 Co-primary endpoint: Success rates at week 12 in the varenicline vs placebo group. Success rates will be defined as Continuous Quit Rate for Weeks 8 to 12 of treatment. Subjects will be classified as responders if they are able to maintain complete abstinence from cigarette smoking in each of the last four study visits (week 9, week 10, week 11, and week 12) with end-expiratory exhaled CO measurements ≤ 10 ppm. This measure will be obtained through reports of cigarette use by means of the Nicotine Use Inventory during the last four study visits (week 9, week 10, week 11, and week 12) confirmed by a measurement of an end-expiratory exhaled carbon monoxide concentration that is ≤ 10 ppm on each study visit Secondary Endpoint: Success rates at week 52 in the varenicline vs placebo group. Success rates will be defined as the Continuous Quit Rate throughout the last three visits (week 24, week 36, and week 44). Subjects will be classified as responders if they are able to maintain abstinence from cigarette smoking during this period of time with end-expiratory exhaled CO measurements ≤ 10 ppm. This measure will be obtained through reports of cigarette use by means of the Nicotine Use Inventory during the last three study visits (week 24, week 36 and week 44) confirmed by a measurement of an end-expiratory exhaled carbon monoxide concentration that is ≤ 10 ppm on each study visit Additional Measures: Given that a better understanding of predictors of smoking cessation can be useful in identifying potential quitters and likely relapsers and that little is known about these predictors in diabetics, the role of different predictors of abstinence at week 24 and at week 52 will also be examined

DETAILED DESCRIPTION:
INTRODUCTION

Cigarette smoking harms nearly every system of the human body, thus causing a broad range of diseases, many of which are fatal. In particular, cardiovascular disease (CVD) is the most important cause of death in those who smoke (1). Both diabetes mellitus and cigarette smoking are well-known risk factors for the development of CVD and atherothrombosis (2,3). It is now acknowledged that endothelial cell dysfunction and clotting activation are not exclusive of diabetes. Cigarette smoking is also associated with functional changes of the endothelium and with an hypercoagulability state (4). It is likely that the combined injurious effects of high blood glucose together with cigarette smoke may be responsible for the observed accelerated course of vascular complications in diabetic patients who smoke.

Findings from both cross-sectional and prospective studies appear to support this notion by consistently showing a heightened risk of morbidity and premature death associated with the development of micro- and macro-vascular disease from the combination of smoking and diabetes. There is evidence that smoking increases the risk of coronary artery disease in type 2 diabetes (5,6). For example, in a prospective cohort of 7,401 female nurses with type 2 diabetes, cigarette smoking was found to be strongly associated with the risk of coronary heart disease (CHD) and this risk increased with the number of cigarettes smoked per day (7). Based on data from 4,540 patients with type 2 diabetes followed in the UK Prospective Diabetes Study (UKPDS), smoking was shown to increase the risk of coronary heart disease in both males and females with type 2 diabetes. The estimated Risk Rate (RR) occurrence of a fatal or non-fatal MI or sudden death attributable to smoking was 1.35 (8). Smoking also increases the risk of stroke (9). Based on patients with type 2 diabetes enrolled in the UKPDS, mathematical models including major confounding variables (including age, sex, atrial fibrillation, etc) estimated that a non-smoking male with a current age of 67 years would have a 6.9% probability of a stroke within 5 years compared with a 10.5% probability for a smoking male of the same age (10). Moreover, several studies have shown that smoking promotes the onset and progression of nephropathy in type 2 diabetes (11-13). In a logistic regression analysis examining associations between gender, age, stage of nephropathy, smoking status, cigarette pack-years, hypertension, total cholesterol, triglycerides, Glycated hemoglobin (HbA1c), and Blood pressure (BP), current and former smoking (P = 0.0012) and number of pack-years (P = 0.011) were shown to be the greatest predictors of the progression of nephropathy (12). Smoking has also been shown to exacerbate markers of kidney failure in this population, such as microalbuminuria (14). In addition, stopping smoking has been shown to reduce the progressive damage to the kidneys in comparison with continued smoking in type 2 diabetes (14).

Because the prevalence of smoking among people with diabetes remains elevated (15), decreasing the exposure to tobacco products is a public health imperative also for subjects with diabetes. Moreover, the most recent US Clinical Guidelines for Treatment of Tobacco Dependence (2008) list diabetes, along with other comorbid medical conditions, as a target group for smoking cessation treatment, due to the increased health risks associated with this disease and smoking (16). It must be also noted that along all known modifiable cardiovascular risk factor (e.g. raised glycemic levels, elevated cholesterol levels, high Body Mass Index) smoking appears to be the most relevant for the reduction of morbidity and mortality in this patient population. Risk management parameters of CVD that include smoking cessation may reduce morbidity and mortality more than tightening glycemic control (17,18).

Surprisingly, there are little data available in the literature on smoking cessation intervention for this specific disease group. Also, no specific information on the efficacy and safety of new pharmacological support for smokers with diabetes can be found. Varenicline is a partial agonist of the α4β2 nicotinic acetylcholine receptor that causes partial stimulation while it competitively inhibits nicotine binding. Recently, randomized, controlled clinical trials have shown that varenicline at a dose of 1 mg twice a day is superior to placebo for smoking cessation (19-21). Varenicline appears to be also more effective than sustained-release bupropion (19). Data from these trials indicate that the most common adverse event attributed to varenicline at a dose of 1 mg twice daily is nausea (19,20). However, the efficacy and safety of varenicline has never been tested in diabetic smokers.

Therefore, the investigators designed a randomized controlled study to test the efficacy and safety of a smoking cessation programme with varenicline tartrate 1 mg BID in diabetic subjects who smoke. The investigators hypothesized that smoking cessation with varenicline could be associated with similar smoking abstinence rates compared to the results obtained in the general population. Given that a better understanding of predictors of smoking cessation (e.g. gender, age at smoking initiation, previous quit attempts, Fagerstrom Test Nicotine Dependence (FTND), motivation, depression, anxiety, social/familial environment, etc.) can be useful in identifying potential quitters and likely relapsers (22) and that little is known about these predictors in diabetics, the role of different predictors of abstinence at the end of the study will also be examined.

STUDY OBJECTIVES This study is intended to assess the safety and efficacy of 12 weeks treatment with varenicline for smoking cessation.

Primary objective: Compare varenicline to placebo for smoking cessation efficacy 12 weeks after treatment (i.e. at week 24) in diabetic smokers

Co-Primary objective: Compare varenicline to placebo for smoking cessation efficacy and safety 1 week after treatment (i.e. at week 13) in diabetic smokers

Secondary objectives: 1) Compare varenicline to placebo for smoking cessation efficacy after treatment at week 52; 2) Compare varenicline to placebo for effects on weight gain in participants successfully quitting smoking; 3) Compare diabetic outcomes in quitters vs relapsers at week 24 and week 52; 4) Examine predictors of abstinence at week 24 and at week 52; 5) Summarize safety data for 12 weeks of treatment with either varenicline or placebo.

METHODS

Study Design The study is a double-blind, placebo-controlled, randomized, clinical trial designed to assess the efficacy and safety of varenicline 1 mg BID in comparison to placebo for smoking cessation in diabetic smokers. The duration of active treatment will be 12 weeks and participants will be followed in the nontreatment phase for an additional 12 weeks (24 week time point). This clinical study has an optional research component to prolong the follow up in the nontreatment phase for a full year (52 week time point). Predictors of abstinence at the end of the study will also be examined.

Study schedule The subjects will have visits in an outpatient clinic setting. The flowcharts in Appendix A and B describe the procedures to be completed at each visit.

Screening visit Activities to be carried out during the screening visit are detailed in the Appendix A. At the screening visit the inclusion/exclusion criteria will be reviewed. The baseline visit will be cancelled if the inclusion/exclusion criteria, including laboratory results, are not met prior to the baseline visit. The baseline visit will occur no less than 3 days and no more than 2 weeks after the screen visit, allowing time for laboratory results to come back.

Baseline visit Activities to be carried out during the baseline visit are detailed in the Appendix A. Inclusion/exclusion criteria will be reviewed once again. At the baseline visit, participants will be instructed on how to prepare to stop smoking and to set a target quit date (TQD), which will be planned to coincide with the Week 1 visit. Also at the baseline visit, each participant will be randomly assigned to either varenicline 1 mg BID + counseling or matched placebo + counseling. Qualified site personnel will dispense the study drug and provide dosing instructions. The participants will be provided approximately. 10 minutes of counseling, in accordance with Agency for Healthcare Research and Quality (AHRQ) guidelines. Diabetic smokers will be subjected to their usual care throughout the study.

Week 1 to 12 visits Subjects will return for visits to the clinic after the baseline visit over the following 12 weeks at Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12. Subsequent to Week 1 Target Quit Date (TQD-visit), visits will occur within 3 days of each scheduled visit date. The subjects will attempt to quit on the target quit date at the Week 1 visit. The quit attempt should occur in the morning prior to the clinic visit that day, so that the subject's last cigarette prior to the quit attempt will be before midnight the night prior to the Week 1 visit. Subjects will be called 3 days after the target quit date (TQD+3) to be reminded of study participation and to receive support for the smoking cessation attempt. These contacts should be no longer than 5 minutes and counselling will follow AHRQ guidelines. Activities to be carried out during these visits are detailed in the Appendix A. At each visit, participants will be provided approximately. 10 minutes of counselling. Study drug will be dispensed by qualified personnel according to the plan illustrated in the Appendix A. Any unused study drug must be returned to the clinic at each visit or upon early termination. All subjects will complete the treatment phase after 12 weeks of participation. Following completion of the Week 12 visit, subjects will continue in the nontreatment follow-up phase of the protocol (see Appendix B). Subjects who do not complete the Week 12 visit will not be eligible to continue. If a subject discontinues study drug prior to the Week 12 visit, the subject may continue study participation as long as they complete the remaining scheduled visits through Week 12. Only subjects completing the week 12 visit will be eligible to continue in the nontreatment follow-up phase of the protocol.

Nontreatment Follow-up (Weeks 13 through 52) Subjects will return for visits to the clinic at Week 24, Week 36, Week 44, and Week 52. Activities to be carried out during these visits are detailed in the Appendix B.

Study Population The study will enroll approximately 150 subjects in each of 2 treatment arms (active drug and matched placebo), for a total of approximately 300 subjects.

STUDY TREATMENTS

Allocation to Study Treatment Diabetic smokers booked for the baseline visit at the smoking cessation center (Centro Per la Prevenzione Cura Tabagimso) will obtain their progressive identification numbers and study drug assignments. Randomization will be performed in permuted blocks of six.

Formulation and Packaging Supplies of varenicline will be in a strength of 0.5 mg tablets and provided in blister cards.

Administration Treatment will begin on the day after the baseline visit. The subjects will take a total of 1 tablet per day for the first 3 days of the dosing period. The dosing will then increase for the next 4 days to 2 tablets per day, 1 in the morning (the first blinded varenicline tablet) and 1 in the evening (the second blinded varenicline tablet). The dosing will then increase to 4 tablets per day, 2 in the morning (the first 2 blinded varenicline tablets) and 2 in the evening (the second 2 blinded varenicline tablets) for the remainder of the study. All subjects are to dose study medication on the day of the Week 1 visit in the morning prior to the visit. DOSING SHOULD OCCUR WITH 240 ML OF WATER AND IT IS RECOMMENDED THAT SUBJECTS EAT PRIOR TO DOSING. There must be at least 8 hours between the morning and evening dosing.

Compliance Subjects will return blister cards at each programmed visit and a dosage record will be recorded.

SAFETY REPORTING

Adverse Events All observed or volunteered adverse events, regardless of treatment group or suspected causal relationship to study drug, will be recorded. This includes symptoms thought to be related to withdrawal from nicotine. Events involving adverse drug reactions, illnesses with onset during the study, or exacerbations of pre-existing illnesses should be recorded. Exacerbation of the disease under study (type 2 diabetes), is defined as a manifestation (sign or symptom) of the illness that indicates a significant increase in the severity of the illness as compared to the severity noted at the start of the trial. It may include worsening or increase in severity of signs or symptoms of the illness, increase in frequency of signs and symptoms of an intermittent illness, or the appearance of a new manifestation/complication. Exacerbation of a pre-existing illness should be considered when a subject requires new or additional concomitant therapy for the treatment of that illness during the trial. In addition, clinically significant changes in physical examination findings and abnormal objective test findings (e.g., laboratory) should also be recorded as adverse events. For all adverse events, the investigator must pursue and obtain information adequate both to determine the outcome of the adverse event and to assess whether it meets the criteria for classification as a serious adverse event. For all adverse events, sufficient information should be obtained by the investigator to determine the causality of the adverse event (i.e., study drug or other illness). The investigator is required to assess causality.

Serious Adverse Events

All serious adverse events (as defined below) regardless of treatment group or suspected relationship to study drug must be reported immediately. A serious adverse event is any adverse drug experience occurring at any dose that:

1. Results in death;
2. Is life-threatening;
3. Results in inpatient hospitalization or prolongation of existing hospitalization;
4. Results in a persistent or significant disability/incapacity.

Any serious adverse event or death must be reported immediately independent of the circumstances or suspected cause if it occurs or comes to the attention of the investigator at any time during the study through 30 days after the last administration of study drug. Any serious adverse event occurring beyond 30 days after the last administration of study drug must be promptly reported if a causal relationship to study drug is suspected.

Clinical Laboratory Parameters and Abnormal Laboratory Test Results

The results of all laboratory tests required by the protocol will be recorded. All clinically important abnormal laboratory tests occurring during the study will be repeated at appropriate intervals until they return either to baseline or to a level deemed acceptable by the investigator or until a diagnosis that explains them is made. The criteria for determining whether an abnormal laboratory test result should be reported as an adverse event are as follows:

1. Test result is associated with accompanying symptoms, and/or
2. Test result requires additional diagnostic testing or medical/surgical intervention, and/or
3. Test result leads to a change in study dosing or discontinuation from the study, significant additional concomitant drug treatment or other therapy, and/or
4. Test result leads to any of the outcomes included in the definition of a serious adverse event, and/or
5. Test result is considered to be an adverse event by the investigator.

The following tests will be completed at the screening and baseline visits: blood chemistry (including sodium, potassium, chloride, BUN, creatinine, glucose, SGOT, SGPT, LDH, alkaline phosphatase, total bilirubin, cholesterol, and triglycerides) and complete blood count. In the event of clinically significant abnormalities, urine samples will be sent for urinalysis. Moreover, the following additional lab tests will be carried out at screening, baseline, week 13, week 24 and week 52 (HbA1c, fasting glucose, total cholesterol, HDL, LDL, triglycerides, insulinemia, albumin to creatinine ratio, and plasma creatinine).

Abnormal Physical Examination Findings Clinically significant changes, in the judgment of the investigator, in physical examination findings (abnormalities) will be recorded as adverse events.

DATA ANALYSIS/STATISTICAL METHODS

Sample Size Determination The sample size calculation for this Randomized Clinical Trial, based on the success quit rates from our previous smoking cessation study (23), indicates that 138 subjects will be required to have 80% power with two-sided 0.05 significance level test to detect a difference of at least 20% quit rate (24 week CQR) between treatment groups. Allowing for a conservative attrition rate of approximately 50%, the target number of participants will be increased to a total of 300.

Methods of Analysis Baseline, demographic and safety data will be listed for all treatment groups. Summary statistics will be provided for each treatment group. The student T-test will be used to compare between mean values of continuous variables in either intervention groups, while the Chi-square test will be used to compare difference between categorical variables. The secondary endpoints will be analyzed using procedures similar to that described above for the primary endpoint. Multivariate logistic regression will be used to identify independent predictors associated with abstinence at week 24 and at week 52.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetic patients (≤ 75 years of age) who are regular smokers (≥10 cigs/day during the past year, with no period of abstinence greater than three months in the past year) and willing to quit.
2. Females of non childbearing potential (surgically sterilized or at least 2 years postmenopausal) who are not nursing may be included. Females of childbearing potential may be included provided that they are not pregnant, not nursing, and are practicing effective contraception.
3. Subjects must be able to be outpatients and be assessed in a clinic setting.
4. Participating subjects must be able to provide written informed consent.

Exclusion Criteria:

1. Subjects currently or within the past 12 months requiring treatment for depression. Subjects with a past or present history of panic disorder, psychosis, or bipolar disorder;
2. Subjects with a current or recent (within the past 12 months) history of alcoholism;
3. Subjects with a requirement to use other medications during the study that might interfere with the evaluation of the study drug (e.g., nicotine replacement therapy);
4. Subjects with a body mass index (BMI) less than 15 or greater than 38, wearing indoor clothing without shoes and determined using the Body Mass Index (BMI);
5. Subjects with evidence or history of clinically significant allergic (except for seasonal allergies at time of dosing), endocrine, gastrointestinal, hematological, hepatic, neurologic, pulmonary, or renal disease or a history of cancer (excluding treated basal cell carcinoma and squamous cell carcinoma). Exceptions to this exclusion may include subjects with a history of mild chronic obstructive pulmonary disease, and stable thyroid disease.
6. Subjects with a history of clinically significant cardiovascular disease. In addition, subjects with uncontrolled hypertension or a screening or baseline systolic blood pressure greater than 160 mm Hg or a diastolic blood pressure greater than 95 mm Hg will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Success rates and safety at week 24 in the varenicline vs placebo. Success rates will be defined as the Continuous Quit Rate since last visit. Maintain abstinence during this period of time with end-expiratory exhaled CO measurements ≤ 10 ppm. | week 24
  Adverse events observed or reported will be recorded. Assessments as to seriousness, severity, and the relationship to treatment and other causes will be made. Physical examination will be performed at the screening visit and at Wk 12. Blood pressure and heart rate will be measured at all visits. BMI and waist will be calculated at the screening visit and at Week 13, 24, 52. Blood chemistry, complete blood count, and urinalysis will be completed at screening, baseline, Week 2 and 12.

SECONDARY OUTCOMES:
Success rates at week 52 in the varenicline vs placebo group. Success rates will be defined as the Continuous Quit Rate (CQR) throughout the last three visits (week 24, week 36, and week 44). | week 52
  Subjects will be classified as responders if they are able to maintain abstinence from cigarette smoking during this period of time with end-expiratory exhaled CO measurements ≤ 10 ppm. This measure will be obtained through reports of cigarette use by means of the Nicotine Use Inventory (NUI) during the last three study visits (week 24, week 36 and week 44) confirmed by a measurement of an end-expiratory exhaled carbon monoxide concentration that is ≤ 10 ppm on each study visit.
"Number of Participants with Adverse Events" | 24-weeks
  Express the percentage of participants with Adverse Events in the active and in the placebo group.
"Change from Baseline in Systolic Blood Pressure" | 24- and 52-weeks
  This measures the % change from baseline. An improvement in systolic blood pressure is anticipated.
"Change from Baseline in HbA1c" | 24- and 52-weeks
  This measures the % change from baseline. An improvement in HbA1c is anticipated
"Change from Baseline in BMI" | 24- and 52-weeks
  This measures the % change from baseline. An slight increase in BMI is expected in the first few months after cessation.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Centro per la Prevenzione e Cura del Tabagimso, Catania, Italy
  - Centro per la Prevenzione eCura del Tabagimso, Catania, Italy

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Russo C, Walicka M, Caponnetto P, Cibella F, Maglia M, Alamo A, Campagna D, Frittitta L, Di Mauro M, Caci G, Krysinski A, Franek E, Polosa R. Efficacy and Safety of Varenicline for Smoking Cessation in Patients With Type 2 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jun 1;5(6):e2217709. doi: 10.1001/jamanetworkopen.2022.17709. PMID 35727580
- [Derived] Russo C, Caponnetto P, Cibella F, Maglia M, Alamo A, Campagna D, Frittitta L, Di Mauro M, Leotta C, Mondati E, Krysinski A, Franek E, Polosa R. A double blind randomized controlled trial investigating efficacy and safety of varenicline for smoking cessation in patients with type 2 diabetes: study protocol. Intern Emerg Med. 2021 Oct;16(7):1823-1839. doi: 10.1007/s11739-021-02684-1. Epub 2021 Mar 18. PMID 33735416